CLINICAL TRIAL: NCT00937378
Title: A Phase III Randomized, Double Blind, Placebo Control, Multicenter Study to Investigate the Efficacy the Efficacy and Safety of SER120 Nasal Spray Formulation in Patients With Nocturia (Non PK Study)
Brief Title: Treatment of Patients With Nocturia (Non-PK Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serenity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPC-SER120-DB2-200902
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2014-04

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SER120 (Experimental)
  Interventions: Drug: SER120
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SER120 — Nasal Spray, once a day
  Arms: SER120
Drug: Placebo — Nasal Spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate a treatment of nocturia. The hypothesis is that SER120 will decrease the number of nocturic episodes compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female 50 years or older
* Nocturia of 6 or more months duration averaging 2 episodes or more per night

Exclusion Criteria:

* CHF
* Diabetes
* Diabetes Insipidus, Renal Insufficiency, Hepatic Insufficiency
* Incontinence
* Illness requiring steroids
* Current or past urologic malignancy
* Nephrotic Syndrome
* Unexplained pelvic masses
* Urinary bladder neurological dysfunction
* Urinary bladder surgery or radiotherapy
* Sleep Apnea
* Pregnant or breast feeding

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Urology Associates, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SER120: All participants received SER120 500 ng once daily for at least 1 week and, if needed, participants were allowed to up-titrate to SER120 750 ng once daily for the remainder of the study.
- Placebo: All participants received placebo once daily for at least 1 week and were allowed to undergo a mock up-titration once daily for the remainder of the study.
Period: Overall Study
Arm/Group | SER120 | Placebo
Started | 167 | 159
Completed | 149 | 141
Not Completed | 18 | 18

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Placebo: All participants received placebo once daily for at least 1 week and were allowed to undergo a mock up-titration on placebo once daily for the remainder of the study.
- Total: Total of all reporting groups
Arm/Group | SER120 | Placebo | Total
Number analyzed (Participants) | 162 | 156 | 318
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (9.1) | 64.6 (8.8) | 64.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 57 | 112
  Male | 107 | 99 | 206
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 152 | 145 | 297
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 162 | 156 | 318

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Nocturic Episodes/Night
Description: Change was calculated as the mean number of nocturic episodes per night between baseline and Week 7
Time Frame: 7 weeks
Population: Intent-to-treat
Measure: Least Squares Mean (Standard Deviation); unit: nocturic episodes per night
Arm/Group | SER120 | Placebo
Number analyzed (Participants) | 162 | 156
nocturic episodes per night | -1.3 (0.8) | -1.2 (0.8)

2. Primary Outcome: Percent of Participants With at Least 50% Decrease in Mean Nocturic Episodes Per Night
Description: Percent of participants achieving at least 50% reduction in nocturic episodes during the last week of treatment compared to baseline
Time Frame: 7 weeks
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | SER120 | Placebo
Number analyzed (Participants) | 162 | 156
Participants | 83 | 64

ADVERSE EVENTS:
Description: Safety Population (only on participants who had received at least one dose of study drug and reported an adverse event).
Arm/Group | SER120 | Placebo
Serious Adverse Events (participants affected / at risk) | 3/167 | 1/159
Other Adverse Events (participants affected / at risk) | 112/167 | 102/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 (N=167) | Placebo (N=159)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Celulitis (Infections and infestations) | 1 (1) | 0 (0)
diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 (N=167) | Placebo (N=159)
Lacrimation increased (Eye disorders) | 11 (11) | 10 (10)
Headache (Nervous system disorders) | 13 (13) | 6 (6)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 53 (53) | 48 (48)
sneezing (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 27 (27)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 16 (16)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes